CLINICAL TRIAL: NCT03743012
Title: Cardiac Rehabilitation Outcomes and Metabolomic Profiles Among Patients With Heart Failure in Western Kenya
Brief Title: Cardiac Rehabilitation and Metabolomics in Heart Failure
Acronym: CROMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Moi Teaching and Referral Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00100126
Record Dates: First submitted 2018-11-14; First posted 2018-11-15 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure
Keywords: rehabilitation; metabolomics
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated cardiac rehabilitation (Experimental): Participants enrolled in integrated cardiac rehabilitation plus usual care
  Interventions: Other: Integrated cardiac rehabilitation
- Usual Care (Active Comparator): Participants receiving usual care only
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Integrated cardiac rehabilitation — Participants enrolled to the integrated cardiac rehabilitation arm will participate in individually tailored rehabilitation sessions that will involve aerobic activity focused on exertion at the participant's aerobic threshold (AT) over a duration of three months.
  Arms: Integrated cardiac rehabilitation
Other: Usual Care — Participants randomized to the usual care arm will be instructed on the benefits of exercise and continue with usual care. Participant activity will be tracked monthly using pedometers for three months of follow up.
  Arms: Usual Care

SUMMARY:
This is a randomized controlled trial of participants with heart failure randomized into usual care plus integrated cardiac rehabilitation or usual care only. The rehabilitation protocol will comprise one month of thrice weekly sessions including supervised aerobic exercises and counseling, followed by two months of monitored home based exercises prescribed weekly.

Cardiopulmonary performance status, depression and quality of life will be assessed at enrollment and upon completion of the protocol using the 6-minute walk time distance test. Plasma samples will be collected and bio-banked for metabolomic profiling and comparative outcome analysis.

DETAILED DESCRIPTION:
Integrated cardiac rehabilitation will comprise one month of thrice weekly sessions of supervised aerobic exercises and counseling, followed by two months of monitored home based exercises prescribed weekly.

Aerobic threshold (AT) will be determined based on perceived rates of exertion as measured using a Borg scale and target heart rate based on Karvonen's formula. Exercise intensity will be prescribed to achieve the earlier of moderate perceived exertion and 50-60% of their maximal target heart rate on a treadmill. Intensity will be increased over the course of the 12 sessions to attain 70-80% of maximal target heart rate. Duration of exercise will also be increased gradually over the 12 sessions in keeping with the study participants perceived rate of exertion.

Participants will be given pedometers and instructed to use these daily for the period of the study. At the end of the first four weeks, the participant's weekly steps will be averaged to establish a baseline weekly step target. Starting in the 4th week,subjects will be instructed to continue exercises at home whilst maintaining a comparable activity level as will be measured by their weekly step counts. Participants will be contacted weekly for the remaining 8 weeks and step targets will be prescribed based on 10% weekly increments.Prior to the start of each exercise session, participants will receive a brief counseling module reflecting the primary goals of cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA Class II or III heart failure
2. Owns a mobile telephone
3. Can participate in supervised exercise three times a week
4. Can read/ primary care giver can read in English or Kiswahili

Exclusion Criteria:

1. Recent acute illness requiring hospitalization in the preceding 4 weeks.
2. Limitation of activity because of factors other than fatigue or exertional dyspnea, such as arthritis, claudication in the legs, angina, advanced co morbidities.
3. Known uncontrolled arrhythmia.
4. Heart failure due to congenital heart disease.
5. Pregnant patients as may be confirmed by patient report or urine pregnancy tests
6. Heart failure due to obstructive cardiomyopathy including mitral stenosis and aortic stenosis.
7. Use of pacemakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
6 minute walk time distance | 3 months
  This study seeks to find out whether 6 minute walk time distance among patients undergoing integrated cardiac rehabilitation is different when compared to usual care study participants.

SECONDARY OUTCOMES:
Depression severity | 3 months
  Change in total depression screening scores using PHQ9 score
Quality of living | 3 months
  Change in quality of living total score as measured by the WHO quality of life scale.

OTHER OUTCOMES:
Metabolomic Profile | 3 months
  This study will secondarily describe pre - post intervention changes in metabolomic profiles in participants with heart failure as measured using mass spectroscopy
Inflammatory Profile | 3 months
  This study will secondarily describe pre - post intervention changes in markers of inflammation such as hsCRP, interleukin-6, TNF-α, and ICAM-1 in participants with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Bloomfield, MD, Principal Investigator — Duke University; Felix Barasa, Principal Investigator — Moi Teaching and Referral Hospital
Locations (1):
- Moi teaching and Referral Hospital, Eldoret, Uasin Gishu County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Feasibility study — https://clinicaltrials.gov/ct2/show/NCT02795936